CLINICAL TRIAL: NCT00790140
Title: Randomized Double Blinded Trial to Investigate Effects of an Enteral Nutritional Supplement Enriched With Eicosapentaenoic Acid on Body Composition,Complications,Stress Response,Immune Function & Quality of Life in After Esophagectomy
Brief Title: Trial of Enteral Nutrition Enriched With Eicosapentaenoic Acid (EPA) in Upper Gastrointestinal Cancer Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Abbott (Industry)
Responsible Party: Professor John V Reynolds, Professor of Surgery, St. James's Hospital, Dublin 8, Ireland
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 900/429/1
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; esophagectomy; enteral feeding; body composition; immunology
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Ensure Plus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immunonutrition Prosure (Active Comparator): This group of patients are to be given a tube feed enriched with 2.2 g Eicosapentaenoic Acid (EPA) per day for 5 days pre surgery and 21 days post surgery
  Interventions: Dietary Supplement: Prosure
- Standard enteral nutrition Ensure Plus (Placebo Comparator): This group are to be given a standard enteral tube feed without EPA for 5 days pre op and 21 days post surgery
  Interventions: Dietary Supplement: Ensure Plus

INTERVENTIONS:
Dietary Supplement: Prosure — This is an enteral tube feed with 125 kcals & 6.65g protein per 100mls. It contains Fat, Carbohydrate, and vitamins and minerals and is enriched with 2.2g Eicosapentaenoic Acid per 500mls of feed. Patients on this trial who are randomized to Prosure will receive the product orally for 5 days prior to surgery and for 21 days post surgery vis a feeding jejunostomy tube
  Other Names: Prosure (Abbott Laboratories)
  Arms: Immunonutrition Prosure
Dietary Supplement: Ensure Plus — This is a standard enteral tube feed with 150 kcals & 6.3 g protein per 100mls as well as carbohydrate, fat and vitamins and minerals. It does not have any active immunonutrients. Patients randomized to this arm will receive the product for 5 days pre op and 21 days post surgery via a feeding jejunostomy tube
  Other Names: Ensure Plus (Abbott Laboratories)
  Arms: Standard enteral nutrition Ensure Plus

SUMMARY:
This study aims to examine whether providing tube feeding with a formula enriched with omega-3 fats is better than traditional standard tube feeding in terms of preserving nutritional status, improving immune function and reducing medical complications following major upper Gut cancer surgery.

DETAILED DESCRIPTION:
Title A double blinded randomized controlled trial to investigate the effects of an enteral nutritional supplement enriched with Eicosapentaenoic acid on long term nutritional status post operatively specifically the maintenance of lean body mass, and its potential impact on quality of life as well as examining the stress response and immune function and in patients undergoing surgical treatment of esophageal cancer.

Investigational medicinal Product(s):

Prosure (Abbott Laboratories)

Comparator:

Ensure Plus (Abbott Laboratories)

Study Objectives To examine whether prolonged supplementation with a nutritional supplement enriched with Eicosapentaenoic acid is superior to standard nutritional products in terms of promoting anabolism and improving quality of life in patients undergoing surgical treatment of esophageal cancer.

Study Design - Prospective randomized controlled trial.

Primary Endpoints:

* Quality of life Scores using EORTC Questionnaires
* Nutritional status on day 21 post oesophagectomy and/or total gastrectomy(specifically lean body mass) and at out patient follow up

Secondary Endpoints:

* Effects on the immuno-inflammatory response to surgery
* Post operative Clinical outcome including SIRS, sepsis and organ failure

ELIGIBILITY:
Inclusion Criteria:

* Adult (male & female) patients >18 years with resectable esophageal cancer

Exclusion Criteria:

* Patients with metastatic disease,
* Non-operable cases,
* Patients requiring chemotherapy/radiotherapy early following surgery,
* Patients with known immunological disorder,
* Emergency esophagectomy cases,
* Patients with cardiac, liver or renal failure,
* Active small intestinal disease eg Crohns disease,
* Allergy to any of the ingredients,
* Uncontrollable Diabetes,
* Use of medications known to affect eicosanoid metabolism in two weeks prior to trial,
* Use of fish oil/n-3 fatty acids,
* Drug Abuse,
* Unable to take preparation for 5 days preoperatively,
* Pregnant women,
* Cessation of enteral feeding for longer than 3 consecutive days post operatively for medical/surgical reasons (e.g. Chyle leaks).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-07; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Preservation of body compostition after surgery | 2 months

SECONDARY OUTCOMES:
Reduced immuno-inflammatory response to surgery | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Healy, BSc RD, Principal Investigator — St. James's Hospital, Dublin 8, Ireland
Locations (1):
- St. James's Hospital,, Dublin, Ireland

REFERENCES:
- [Derived] Healy LA, Ryan A, Doyle SL, Ni Bhuachalla EB, Cushen S, Segurado R, Murphy T, Ravi N, Donohoe CL, Reynolds JV. Does Prolonged Enteral Feeding With Supplemental Omega-3 Fatty Acids Impact on Recovery Post-esophagectomy: Results of a Randomized Double-Blind Trial. Ann Surg. 2017 Nov;266(5):720-728. doi: 10.1097/SLA.0000000000002390. PMID 28742713
- [Derived] Ryan AM, Reynolds JV, Healy L, Byrne M, Moore J, Brannelly N, McHugh A, McCormack D, Flood P. Enteral nutrition enriched with eicosapentaenoic acid (EPA) preserves lean body mass following esophageal cancer surgery: results of a double-blinded randomized controlled trial. Ann Surg. 2009 Mar;249(3):355-63. doi: 10.1097/SLA.0b013e31819a4789. PMID 19247018